CLINICAL TRIAL: NCT07228637
Title: Pursuing Exploration Into the Supportive Care Needs and Intervention Preferences of Survivors of Testicular Cancer (PERSIST): A Mixed Methods Pilot Study
Brief Title: Pursuing Exploration Into the Supportive Care Needs and Intervention Preferences of Survivors of Testicular Cancer
Acronym: PERSIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shelley Johns, Associate Professor of Medicine and Walther Scholar in Psycho-Oncology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22340
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Testicular Cancer
Keywords: Fear of Cancer Recurrence; Anxiety; Acceptance and Commitment Therapy; Supportive Care Needs
MeSH Terms: conditions — Testicular Neoplasms; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants (N = 70) will be randomly assigned in equal numbers to the ACT-based coaching program or an education/support coaching program using a stratified block randomization scheme to balance the groups by patient-reported time since treatment completion (last testicular cancer treatment was less than 2 years ago vs. last testicular cancer treatment was 2-5 years ago).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching Program 1: Acceptance and Commitment Therapy (ACT) (Experimental): Testicular cancer survivors in the ACT-based coaching arm will learn new and more adaptive ways to respond to fear of cancer recurrence and other difficult internal experiences (e.g., thoughts, feelings, body sensations).
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) Coaching
- Coaching Program 2: Education and Support (Active Comparator): Testicular cancer survivors in the education and support coaching arm will discuss their cancer-related concerns and receive education on supportive services and resources available locally and nationally.
  Interventions: Behavioral: Education and Support Coaching

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) Coaching — Across six weekly 90-minute online group sessions, testicular cancer survivors in the ACT coaching arm will practice various mindfulness exercises, clarify their values, and set specific values-based action goals in alignment with their values. Through in-session and home practice of skills, participants learn new and more adaptive ways to respond to fear of cancer recurrence and other difficult internal experiences (e.g., thoughts, feelings, body sensations). Participants receive handouts on session topics and a link to guided mindfulness practices developed by our team. Participants will be asked to track their home practices on provided logs.
  Arms: Coaching Program 1: Acceptance and Commitment Therapy (ACT)
Behavioral: Education and Support Coaching — Across six weekly 90-minute sessions, testicular cancer survivors in the education and support coaching arm are directed to resources for practical support, health information, and contact information for available community and national resources and support. Sessions include an orientation to testicular cancer survivorship and recurrence risks, education regarding common quality-of-life concerns experienced by cancer survivors, and an overview of community and national resources for addressing these concerns. Participants receive handouts summarizing session topics and are asked to review them as homework.
  Arms: Coaching Program 2: Education and Support

SUMMARY:
This trial tests the impact of an Acceptance and Commitment Therapy (ACT)-based coaching program delivered via videoconferencing on fear of cancer recurrence (primary outcome), anxiety, other symptoms, health-related quality of life, and coping (secondary outcomes) in survivors of testicular cancer. ACT includes experiential training in present moment awareness (e.g., mindfulness meditation, performing activities with greater awareness), coping adaptively with difficult internal experiences (e.g., thoughts, feelings, body sensation), identifying personally meaningful values, and pursuing activities consistent with these values. Testicular cancer survivors (N=70) will be randomly assigned in equal numbers to either an ACT-based coaching program or an education/support coaching program, both delivered via videoconferencing. Survivors in both conditions will participate in six weekly 90-minute online group sessions. Outcomes will be assessed at baseline, 2 weeks post-intervention, and 3 months post-intervention. The investigators hypothesize that ACT will lead to improved primary and secondary outcomes as compared to education/support. Study findings will inform a large-scale trial of intervention efficacy.

DETAILED DESCRIPTION:
This trial evaluates the feasibility, acceptability, and preliminary efficacy of an Acceptance and Commitment Therapy (ACT)-based coaching program delivered via videoconferencing on fear of cancer recurrence (primary outcome), anxiety, other symptoms, health-related quality of life, and coping (secondary outcomes) in survivors of testicular cancer. The study team is recruiting testicular cancer survivors who have received care at the Indiana University Simon Comprehensive Cancer Center. Potentially eligible patients will be mailed an introductory letter signed by their oncologist and the PI along with a consent form and study flyer. The letter has a number to call if they did not wish to be contacted further. A research assistant (RA) will call all prospective participants who do not opt out approximately 1 week after the letter was mailed. The RA will describe the study as outlined in the consent form and answer any questions. Then the RA will administer an eligibility screening to interested patients. Eligible and interested patients will provide verbal consent before completing a baseline assessment online. Following baseline assessments, patients (N = 70) will be randomly assigned in equal numbers to the ACT-based coaching program or an education/support coaching program using a stratified block randomization scheme to balance the groups by patient-reported time since treatment (last testicular cancer treatment was less than 2 years ago vs. last testicular cancer treatment was 2-5 years ago). Patients in both study conditions will complete six weekly 90-minute group sessions via videoconferencing, with the first session occurring within three weeks of baseline. For both conditions, participants will log their adherence to home practice assignments between sessions. Feasibility will be examined via accrual, attrition, and adherence rates, and acceptability will be evaluated using a mixed methods approach (quantitative and qualitative).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed with testicular cancer (any type, stage, or risk category) without evidence of active distant disease at time of study entry
* Completed surgery, chemotherapy, radiation therapy, and/or stem cell transplant 5 years or less prior to enrollment
* Willing to provide authorization to be contacted by email
* Willing to complete surveys
* Willing to participate in six, 90-minute intervention sessions
* Able to speak and read English
* Has clinically significant fear of cancer recurrence (FCR-4 score = 9 or higher) and/or anxiety (GAD-2 score = 3 or higher) at eligibility screening

Exclusion Criteria:

* Completed surgery, chemotherapy, radiation therapy, and/or stem cell transplant less than 2 weeks prior to enrollment (excluding to avoid acute toxicity side effects of treatment)
* Patient has co-morbidities or deficits that would impair participation in the study, including:

  1. history of neurological disorder or traumatic brain injury (e.g., stroke, encephalitis, epilepsy, loss of consciousness greater than 10 minutes);
  2. severe depressive symptoms (PHQ-2 score = 5 or higher at screening),
  3. active substance abuse or uncontrolled bipolar disorder, schizophrenia, or psychosis;
  4. obvious hearing and/or communicative disability that would impair their participation
* Patient is currently participating in "The Platinum Study" (PI: Lois Travis)
* Currently participating in psychotherapy focused on cancer-specific adjustment/support
* Currently participating in any behavioral/psychosocial research study that has the potential to skew results of this study or the study in which the survivor is participating

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Scale - 7 items (FCR-7) | 2 weeks and 3 months post-intervention
  This 7-item measure includes 6 items assessing feelings associated with cancer recurrence and cognitive and behavioral responses to fear of cancer recurrence on 5-point scales (1=not at all to 5=all the time). Question 7 is a single item assessing the extent to which fear of cancer recurrence intrudes on thoughts and activities on a 0-10 scale (0=not at all to 10=a great deal). The 7 items are summed with higher total scores indicating greater fear of cancer recurrence. The total score range is from 6 to 40. This is the primary outcome measure.

SECONDARY OUTCOMES:
Fear of Cancer Recurrence Inventory (FCRI) | 2 weeks and 3 months post-intervention
  This 42-item measure includes items assessing fear of cancer recurrence-related triggers (8 items), severity (9 items), psychological distress (4 items), functioning impairment (6 items), insight (3 items), reassurance seeking (3 items), and coping strategies (9 items). Items are rated on 5-point scales (0=never/not at all to 4=all the time/a great deal) to indicate the extent to which participants have felt fearful during the past month. Item #13 is reverse-scored and then the 42 items are summed with higher total scores indicating greater fear of cancer recurrence. The total score range is 0 to 168. This is a secondary outcome measure.
Fear of Cancer Recurrence Global Improvement | 2 weeks and 3 months post-intervention
  This retrospective global rating of improvement in fear of cancer recurrence provides a patient-centered approach to assessing change that is clinically meaningful. At each post-intervention time points, participants are asked, "Overall, since starting the study program, would you say that your fear of recurrence is: worse, about the same, or better?" Those reporting their fear of cancer recurrence as "better" are then asked if their fear is "a little better, somewhat better, moderately better, a lot better, or completely better." Responses are coded on a 7-point scale such that 0=worse, 1=about the same, 2=a little better, 3=somewhat better, 4=moderately better, 5=a lot better, and 6=completely better, with a higher score indicating greater improvement in fear of cancer recurrence since starting the study program to which they were randomly assigned. This is a secondary outcome measure.
Generalized Anxiety Disorder Scale - 7 items (GAD-7) | 2 weeks and 3 months post-intervention
  Seven items are rated on 4-point scales (0=not at all to 3=nearly every day) to indicate how often in the past 2 weeks participants have been bothered by symptoms of anxiety. The 7 items are summed with higher total scores indicating greater anxiety. The total score range is 0 to 21. This is a secondary outcome measure.
Patient Health Questionnaire - 8 items (PHQ-8) | 2 weeks and 3 months post-intervention
  Seven items are rated on 4-point scales (0=not at all to 3=nearly every day) to indicate how often in the past 2 weeks participants have been bothered by symptoms of anxiety. The 7 items are summed with higher total scores indicating greater anxiety. The total score range is 0 to 21. This is a secondary outcome measure.
Impact of Events Scale-Revised (IES-R) | 2 weeks and 3 months post-intervention
  Twenty-two items are rated on 5-point scales (0=not at all to 4=extremely) to indicate how often in the past 7 days participants have been bothered by post-traumatic stress symptoms, including experiences of intrusion, avoidance, and hyperarousal. The 22 items are summed with higher total scores indicating greater post-traumatic stress. The total score range is 0 to 88. This is a secondary outcome measure.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health | 2 weeks and 3 months post-intervention
  This 10-item measure assesses global health, including physical, mental, and social well-being. With the exception of pain, which is rated on a 0 to 10 scale, all items are rated on 5-point scales from 1 to 5. The item on pain is recoded from a 0-10 to a 1-5 scale and reverse scored. Two additional items are reverse scored. Four of the items are summed, with higher physical quality of life subscale scores indicating better physical quality of life. Four other items are also summed with higher psychological quality of life subscale scores indicating better psychological quality of life. The subscale scores are converted to T-scores with a range from 16.2 to 67.7 for physical quality of life and a range from 21.2 to 67.6 for psychological quality of life. Higher T-scores for the physical and psychological quality of life subscales indicate a better outcome. The population mean for T-scores is 50 with a standard deviation of 10. This is a secondary outcome measure.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (4a) | 2 weeks and 3 months post-intervention
  This 4-item measure assesses the perceived interference of pain with functioning in several life domains in the past 7 days. Each item is rated on a 5-point scale (1=not at all to 5=very much). The 4 items are summed with higher total scores indicating greater pain-related interference. The total scores are converted to T-scores with a range from 41.6 to 75.6. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (4a) | 2 weeks and 3 months post-intervention
  This 4-item measure assesses perceived fatigue severity in the past 7 days. Each item is rated on a 5-point scale (1=not at all to 5=very much). The 4 items are summed with higher total scores indicating greater fatigue severity. The total scores are converted to T-scores with a range from 33.7 to 75.8. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (4a) | 2 weeks and 3 months post-intervention
  This 4-item measure assesses perceived sleep disturbance in the past 7 days. Each item is rated on a 5-point scale (1=not at all/very good to 5=very much/very poor). Two items (Sleep109, Sleep116) are reverse scored. The 4 items are summed with higher total scores indicating greater sleep disturbance. The total scores are converted to T-scores with a range from 32.0 to 73.3. Higher T-scores indicate a worse outcome. The population mean for T-scores is 50 with a standard deviation of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function (4a) | 2 weeks and 3 months post-intervention
  This 4-item measure assesses perceived cognitive functioning in the past 7 days. Each item is rated on a 5-point scale (1=very often/several times a day to 5=never). The 4 items are summed with higher total scores indicating better cognitive functioning. The total scores are converted to T-scores with a range from 24.99 to 61.13. Higher T-scores indicate a better outcome. The population mean for T-scores is 50 with a standard deviation of 10.
Multidimensional Psychological Flexibility Inventory (MPFI) | 2 weeks and 3 months post-intervention
  Thirty-five items from the Multidimensional Psychological Flexibility Inventory are being used to assess one aspect of psychological flexibility (i.e., acceptance; 5 items) and six aspects of psychological inflexibility (i.e., experiential avoidance, cognitive fusion, lack of contact with the present moment, attachment to the conceptualized self, lack of values clarity, and inaction; 30 items total). Across items, participants rate their behavior on 6-point scales from 1=never true to 6=always true. Separate mean scores across the 5 acceptance items and the 30 psychological inflexibility items are calculated, with mean scores ranging from 1 to 6 on each. Higher mean scores reflect greater acceptance and psychological inflexibility, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A. Johns, PsyD, Principal Investigator — Indiana University
Locations (1):
- Indiana University - Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of this trial will be presented at professional meetings and published in peer-reviewed journals. The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. The data set will contain necessary identifiers, excluding those prohibited by HIPAA. The investigators will be required to sign a data use agreement and obtain Institutional Review Board (IRB) approval before receiving the data set.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data set will be made available to qualified investigators within 6 months of the publication of the primary outcome paper. Data will be available for at least 6 years.
Access Criteria: The data set and supporting information will be made available to qualified investigators to allow replication of analyses or secondary data analyses. The PI will review requests for data access. The investigators will be required to sign a data use agreement and obtain IRB approval before receiving the data set. The mechanism for data sharing will be reviewed by the IRB.